CLINICAL TRIAL: NCT05050734
Title: A Randomized Waitlist-Controlled Pilot Trial of Online-Delivered Comprehensive Behavioral Intervention for Tics-Enhanced (CBIT-E)
Brief Title: Online-Delivered Comprehensive Behavioral Intervention for Tics-Enhanced (CBIT-E)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marquette University (Other)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HR-3837
Record Dates: First submitted 2021-09-03; First posted 2021-09-20 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Persistent Tic Disorders; Tourette Disorder
Keywords: Persistent Tic Disorders; Tourette Disorder; Tics; Behavior Therapy; Children
MeSH Terms: conditions — Tourette Syndrome; Tics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBIT-E (Experimental): For those randomized to CBIT-E, treatment will be administered according to the standard CBIT manual, which includes psychoeducation, functional assessment/interventions, habit reversal training, relaxation techniques, and a motivational reward program. However, there will be two modifications. CBIT-E will include additional in-session and out of session practice of exercises, called competing response. Treatment will include a screening visit, baseline assessment, 11 weeks (9 sessions) of CBIT-E, a post treatment assessment, and a three-month follow up assessment. Further, starting after session 3, there will be four 15-minute practice periods scheduled each week between sessions. During these practice periods, the child and therapist will meet over Microsoft Teams and the therapist will administer an enhanced reward task.
  Interventions: Behavioral: Comprehensive Behavioral Intervention for Tics - Enhanced (CBIT-E)
- Waitlist Control (WLC) (No Intervention): These participants will not receive treatment during the 11-week period. Instead, they will be placed on a waitlist to receive standard CBIT following the end of the study period. The final assessment will be approximately 11 weeks after baseline.

INTERVENTIONS:
Behavioral: Comprehensive Behavioral Intervention for Tics - Enhanced (CBIT-E) — Behavioral treatment for persistent tic disorders.
  Arms: CBIT-E

SUMMARY:
The purpose of this pilot trial is to examine the preliminary efficacy of online-delivered Comprehensive Behavioral Intervention for Tics - Enhanced (CBIT-E). In the study, 30 children with persistent tic disorders (PTDs) will be recruited via information provided to patients of the Marquette University (MU) Tic Disorders Specialty Clinic (TDSC) and information conveyed via local medical health professionals, with the goal of randomizing 10 participants to each group. For those randomized to CBIT-E, treatment will be administered according to the standard CBIT manual, but there will be two modifications. CBIT typically consists of the implementation of strategies to help manage the environment related to tics and the implementation of an exercise to engage in when an individual feels the urge to tic. CBIT-E will include these same techniques, plus additional in-session and out of session practice of the exercises, called competing responses, that individuals use when they feel the urge to tic. Treatment will be delivered over Microsoft Teams, which is a secure video conferencing system. The therapist will administer treatment from a private room in the Marquette University Tic Disorder Specialty Clinic, while the parent and child will be at their home. Treatment will include a screening visit, baseline assessment, 11 weeks (9 sessions) of CBIT-E, a post treatment assessment, and a three-month follow up assessment. Further, starting after session 3, there will be four 15-minute practice periods scheduled each week between sessions. During these practice periods, the child and therapist will meet over Microsoft Teams and the therapist will administer an enhanced reward task.

Children randomized to the waitlist control (WLC) will not receive treatment during the 11-week period. Instead, they will be placed on a waitlist to receive standard CBIT following the end of the study period. Participants in this group will complete a screening visit, baseline assessment, and a final assessment, which will occur approximately 11 weeks after baseline.

ELIGIBILITY:
Inclusion Criteria:

* ages 9-17
* meets Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) diagnostic criteria for TD or PTD
* at screening visit, a Parent Tic Questionnaire (PTQ) total score > 18 and < 60 OR > 12 and < 40 if persistent tic disorder (for total scores > 60 on the PTQ, the research team will examine the patient's global functioning to determine participation appropriateness. The research team will consider if other treatments, such as medication, may be more appropriate for participants with PTQ total scores > 60. If the participant is already taking tic medication, or tic medication has been unsuccessful in the past, then he/she may be considered for the study)
* at baseline visit, a Yale Global Tic Severity Score (YGTSS Total Score) > 14 and < 30 OR > 10 and < 20 if persistent tic disorder (for total scores > 30 on the YGTSS, the research team will examine the patient's global functioning to determine participation appropriateness)
* no history of behavioral treatment for tics, including self-guided therapy programs for tics
* unmedicated or on stable medication for tics and other psychiatric disorder for at least 6 weeks, with no planned changes during study participation
* access to a personal computer (desktop or laptop) with a camera
* access to an Internet connection with a minimum speed of 5 megabytes per second (Mbps)
* fluent English speaker.

Exclusion Criteria:

* co-occurring disorders that require more immediate treatment or change to current treatment
* T-Score < 37 on the Wechsler Abbreviated Scale of Intelligence (WASI) - Vocabulary subtest
* T-Score > 70 on the inattention or hyperactivity/impulsivity scales of the Conners 3-Parent Short (C 3-PS).

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale (YGTSS) | Change from baseline at post-treatment (11 weeks after baseline) and change from post at follow-up (3 months after post)
  Clinician-rated measure that assesses motor and vocal tic severity and impairment over the past week. Motor and vocal tic number, frequency, intensity, complexity, and interference are rated on a 0-5 scale and summed to create separate motor and vocal tic severity scores (each ranging from 0-25). These ratings are combined to create a total tic severity score (Range = 0-50). Clinicians also rate overall tic-related impairment on a 50-point scale. Higher scores are related to more tic severity/impairment.

SECONDARY OUTCOMES:
Clinical Global Impression-Improvement (CGI-I) Scale | Will be completed by the independent evaluator at post (11 weeks after baseline) and 3-month follow-up (3 months after post)
  Clinician-rated scale used to assess overall treatment response. Ratings on the CGI-I range from 1 (very much improved) to 8 (very much worse). CGI-I scores of 2 (much improved) or 1 (very much improved) indicate positive treatment response. Higher scores are related to worse treatment response.

CONTACTS AND LOCATIONS:
Locations (1):
- Marquette University, Milwaukee, Wisconsin, United States